CLINICAL TRIAL: NCT01031446
Title: A Phase Ib/II Study of Cisplatin, Paclitaxel, and RAD001 in Patients With Metastatic Breast Cancer
Brief Title: Cisplatin, Paclitaxel, and Everolimus in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ingrid Mayer, MD, Assistant Professor of Medicine; Clinical Director, Breast Cancer Program, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 0949; P30CA068485 (NIH); VU-VICC-BRE-0949; IRB# 090673
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; Human epidermal growth factor (HER2)-negative breast cancer; triple-negative breast cancer; hormone-resistant breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Cisplatin; Everolimus; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: cisplatin; Drug: everolimus; Drug: paclitaxel; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cisplatin — Given through a vein in the arm 1 time a week for 3 weeks, then a one week break and then begin the process again.
Drug: everolimus — Taken daily by mouth.
Drug: paclitaxel — Given through a vein in the arm 1 time a week for 3 weeks, then a one week break and then begin the process again.
Other: laboratory biomarker analysis — Blood collection

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving cisplatin and paclitaxel together with everolimus may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects of giving cisplatin and paclitaxel together with everolimus and to see how well it works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Safety profile of cisplatin, paclitaxel, and everolimus (RAD001) in patients with metastatic breast cancer. (Phase I)
* Progression-free survival (Phase II)

Secondary

* Overall response rate
* Time to progression
* Number of patients with worst-grade toxicities Tertiary
* To determine p53, p63, p73, and phosphatase and tensin homolog (PTEN) levels by immunohistochemistry (IHC).
* To screen for exon 9 (E542K and E545K), exon 20 (H1047R), and phosphatidylinositol 3-kinase (PI3K) (p110α) mutations in DNA extracted from paraffin blocks.
* To correlate IHC results with clinical outcome and with the different subtypes of breast cancer determined by molecular classification (basal-type vs luminal A vs luminal B) based on microarrays of RNA extracted from formalin-fixed paraffin-embedded blocks.
* To generate microarrays of RNA extracted from fresh-frozen core biopsies (when available) to identify a pretreatment gene signature that mirrors the established p63 and p73 gene signatures that predict response to treatment.

OUTLINE: This is a multicenter study.

Patients receive oral everolimus once daily on days 1-28 and cisplatin IV over 1 hour and paclitaxel IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Tumor tissue samples are collected at baseline for correlative studies.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive mammary carcinoma

  * Stage IV disease
  * Basal-like disease (triple-negative, hormone-refractory, HER2-negative)
* No locally recurrent breast cancer
* No symptomatic brain metastases

  * Patients with a history of brain metastases are eligible provided they are clinically stable for > 3 weeks after completion of radiotherapy and are not taking steroids or therapeutic anticonvulsants that are cytochrome P450 3A4 (CYP3A4) modifiers
  * Patients with asymptomatic brain metastases are eligible provided they are not taking prophylactic anticonvulsants that are CYP3A4 modifiers

PATIENT CHARACTERISTICS:

* Pre- or post-menopausal
* European Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy ≥ 6 months
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 times ULN (≤ 3 times ULN in the presence of liver metastasis)

  * Direct bilirubin will be measured in patients with Gilbert syndrome
* serum glutamate oxaloacetate transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) ≤ 1.5 times ULN (≤ 3 times ULN in the presence of liver metastasis)
* Alkaline phosphatase ≤ 3 times ULN (in the presence of liver metastasis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment
* Able to swallow and retain oral medication
* No malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection requiring parenteral antibiotics
  * Impaired lung function (chronic obstructive pulmonary disease or lung conditions requiring oxygen therapy)
  * New York Heart Association class III-IV congestive heart failure
  * Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within the past 6 months
  * Uncontrolled hypertension (systolic BP > 180 mm Hg or diastolic BP > 100 mm Hg, found on 2 consecutive measurements separated by a 1-week period and despite adequate medical support)
  * Clinically significant cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment [grade 3 according to NCI Common Toxicity Criteria for Adverse Events v3.0])
  * Uncontrolled diabetes (hyperosmolar state, ketoacidosis, etc.)
  * Psychiatric illness or social situations that would compromise patient safety or limit compliance with study requirements including maintenance of a compliance/pill diary
* No symptomatic neuropathy ≥ grade 2
* No other invasive cancer within the past 5 years except for completely resected basal cell or squamous cell carcinoma of the skin or successfully treated cervical carcinoma in situ
* No hypersensitivity to paclitaxel or drugs using the vehicle Cremophor, Chinese hamster ovary cell products, or other recombinant human antibodies
* No history of hepatitis B or C

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* Prior total cumulative life-time dose of doxorubicin ≤ 360 mg/m^2 or epirubicin ≤ 640 mg/m^2
* No more than 4 prior chemotherapy treatments in the metastatic setting (not including endocrine therapy or single-agent biologic therapy)
* At least 2 weeks since prior investigational drugs
* At least 14 days since prior and no concurrent herbal or dietary supplements
* At least 14 days since prior and no concurrent CYP3A4 inducers
* At least 7 days since prior and no concurrent CYP3A4 inhibitors
* Concurrent radiotherapy to painful bone metastases or areas of impending bone fracture allowed provided radiotherapy is initiated before study entry
* No other concurrent anticancer therapy (chemotherapy, radiotherapy, surgery, immunotherapy, hormonal therapy, biologic therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Mayer, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Erlanger Cancer Center at Erlanger Hospital - Baroness, Chattanooga, Tennessee
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Regional Cancer Center at Baptist Riverside, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to accrual in October 2009 and ran to June 2011.
Pre-assignment Details: Fifty-seven patients consented for this study, two were determined ineligible to participate.
Groups:
- RAD001 and Cisplatin and Pacletaxel: RAD001 (Everolimus) by mouth once a day. Cisplatin intravenously (IV) weekly for 3 weeks, then 1 week of rest; paclitaxel IV weekly for 3 weeks, then 1 week of rest. One cycle = 4 weeks. All patients began at the same dose level of the study drugs with no de-escalation of dose, thus results for Phase I and II were combined
Period: Overall Study
Arm/Group | RAD001 and Cisplatin and Pacletaxel
Started | 55
Completed | 0
Not Completed | 55
Not completed — Disease Progression | 38
Not completed — Adverse Event | 9
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 3
Not completed — Still on treatment | 1

BASELINE CHARACTERISTICS:
Groups:
- RAD001 Cisplatin Paclitaxel: RAD001 (Everolimus) by mouth once a day. Cisplatin intravenously (IV) weekly for 3 weeks, then 1 week of rest; paclitaxel IV weekly for 3 weeks, then 1 week of rest. One cycle = 4 weeks.
Arm/Group | RAD001 Cisplatin Paclitaxel
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Maximum Feasible Dose in Milligrams Per Meter Squared of Body Surface Area (mg/m2) of Cisplatin and Paclitaxel for Women With Metastatic Breast Cancer
Description: The recommended dose for the Phase II trial will be the most prevalent dose delivered per week in Phase I that allows for safe and feasible administration of the medications.The maximum tolerated dose (MTD) is defined as the dose preceding that at which 2 or more of 3 patients experience dose-limiting toxicity (DLT) during the initial cycle of therapy. DLTs include Common Toxicity Criteria (CTC) Grade 4 neutropenia (absolute neutrophil count [ANC] < 0.5 x 10 9/L for > 5 days), febrile neutropenia (ANC < 1.0 x 10 0/L with fever > 38.5 degrees Centigrade) or documented infection associated with Grade 3-4 neutropenia, CTC Grade 4 thrombocytopenia < 25 x 10 9/L or CTC Grade 3 < 50-25 x 10 9/L thrombocytopenia with bleeding, and Grade 3-4 non-hematologic toxicity despite symptomatic therapy.
Time Frame: at 8 weeks
Population: Patients enrolled to determine the safety profile and recommended doses of cisplatin + paclitaxel + everolimus (RAD001) in women with metastatic breast cancer
Measure: Number; unit: mg/m2
Groups:
- RAD001 and Cisplatin and Paclitazel: Cisplatin intravenously (IV) weekly for 3 weeks, then 1 week of rest; paclitaxel IV weekly for 3 weeks, then 1 week of rest. Everolimus (RAD001) po daily. One cycle = 4 weeks
Arm/Group | RAD001 and Cisplatin and Paclitazel
Number analyzed (Participants) | 3
mg/m2
  Cisplatin | 25
  Paclitaxel | 80

2. Primary Outcome: Maximum Feasible Dose in mg of RAD001 (Everolimus)for Women With Metastatic Breast Cancer
Description: The recommended dose for the Phase II trial will be the most prevalent dose delivered per day in Phase I that allows for safe and feasible administration the medication. The MTD is defined as the dose preceding that at which 2 or more of 3 patients experience dose-limiting toxicity (DLT) during the initial cycle of therapy. DLTs include Common Toxicity Criteria (CTC) Grade 4 neutropenia (absolute neutrophil count [ANC] < 0.5 x 10 9/L for > 5 days), febrile neutropenia (ANC < 1.0 x 10 0/L with fever > 38.5 degrees Centigrade) or documented infection associated with Grade 3-4 neutropenia, CTC Grade 4 thrombocytopenia < 25 x 10 9/L or CTC Grade 3 < 50-25 x 10 9/L thrombocytopenia with bleeding, and Grade 3-4 non-hematologic toxicity despite symptomatic therapy
Time Frame: at 8 weeks
Population: Patients enrolled to determine the safety profile and recommended dose of cisplatin + RAD001 + paclitaxel in women with metastatic breast cancer
Measure: Number; unit: mg
Groups:
- RAD001 and Cisplatin and Paclitaxel: Cisplatin intravenously (IV) weekly for 3 weeks, then 1 week of rest; paclitaxel IV weekly for 3 weeks, then 1 week of rest. Everolimus (RAD001) po daily. One cycle = 4 weeks
Arm/Group | RAD001 and Cisplatin and Paclitaxel
Number analyzed (Participants) | 3
mg | 5

3. Secondary Outcome: Patients With Overall Response
Description: Per Response Evaluation Criteria in Solid Tumor (RECIST) criteria v. 1.0: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions
Time Frame: every 12 weeks
Population: Patients for whom an overall response could be measured. Four patients were not evaluable due to: withdrew after beginning treatment (1) and not evaluable due to only 1 cycle of treatment (3).
Measure: Number; unit: participants
Groups:
- RAD001 and Cisplatin and Paclitaxel: Patients receive cisplatin IV 25 mg/m2, paclitaxel IV 80 mg/m2 (both drugs once weekly for 3 weeks followed by 1 week of rest), and RAD001 5 mg by mouth daily. 1 cycle = 4 weeks.
Arm/Group | RAD001 and Cisplatin and Paclitaxel
Number analyzed (Participants) | 51
participants
  Complete Response | 1
  Partial Response | 12
  Progressive Disease | 11
  Stable Disease | 27

4. Secondary Outcome: Time to Progression
Description: Duration in months from date on-study to date patient exhibited progressive disease
Time Frame: Up to 64 weeks
Population: Patients who were available for determination of duration of time to progressive disease. Time to progression is unknown for 8 Phase II patients due to: on-treatment (1), toxicity (3), withdrew after beginning treatment (1), and no progression (3)
Measure: Median (Full Range); unit: months
Arm/Group | RAD001 and Cisplatin and Paclitaxel
Number analyzed (Participants) | 47
months | 4.0 [0.4 to 23.0]

5. Primary Outcome: Patients With Progression-free Survival
Description: Patients who had not experienced disease progression and who were alive at 6 months after study entry
Time Frame: at 6 months
Population: Patient who received the study drugs. Four patients were not available for measurement of progression at 6 months: toxicity (3), withdrew after beginning treatment (1)
Measure: Number; unit: participants
Arm/Group | RAD001 and Cisplatin and Paclitaxel
Number analyzed (Participants) | 51
participants | 21 [0 to 23]

6. Secondary Outcome: Time to Progression in Patients With Metastatic Basal-like Breast Cancer.
Description: Median duration in months from on-study to disease progression in patients with metastatic basal-like breast cancer. All patients with basal-like breast cancer are negative for estrogen, progesterone, and human epidermal growth factor (HER2) receptors.
Time Frame: Up to 64 weeks
Population: Patients who are negative for estrogen, progesterone and HER2 receptors. Time to progression was not determined for 5 patients in this group: toxicity (2), withdrew after beginning treatment (1), no progression (1), and on-treatment (1).
Measure: Median (Full Range); unit: months
Arm/Group | RAD001 and Cisplatin and Paclitaxel
Number analyzed (Participants) | 31
months | 4.0 [0.4 to 23.0]

ADVERSE EVENTS:
Groups:
- RAD001 and Cisplatin and Paclitaxel: RAD001 (Everolimus) by mouth once a day. Cisplatin intravenously (IV) weekly for 3 weeks, then 1 week of rest; paclitaxel IV weekly for 3 weeks, then 1 week of rest. One cycle = 4 weeks.
Arm/Group | RAD001 and Cisplatin and Paclitaxel
Serious Adverse Events (participants affected / at risk) | 9/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 and Cisplatin and Paclitaxel (N=55)
pain-abdomen (Gastrointestinal disorders) | 3 (6)
death not associated with CTCAE term-disease progression NOS (General disorders) | 3 (3)
Left maxillary odontogenic abscess and cellulitis (Infections and infestations) | 1 (1)
glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (2)
pain-back (Musculoskeletal and connective tissue disorders) | 2 (3)
neutrophils (Blood and lymphatic system disorders) | 2 (4)
leukocytes (Blood and lymphatic system disorders) | 1 (2)
platelets (Blood and lymphatic system disorders) | 1 (2)
cholecystitis (Hepatobiliary disorders) | 1 (2)
malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
infection with unknown ANC-mucosititis (Infections and infestations) | 1 (1)
infection with unknown ANC-wound, methicillin-resistant Staphylococcus aureus (Infections and infestations) | 1 (1)
febrile neutropenia, ANC < 1.0 x 10e9L, fever ≥ 38.5 degrees Celsius (Blood and lymphatic system disorders) | 1 (1)
fever in absence of neutropenia w/ neutropenia defined as ANC < 1.0 x 10e9L (General disorders) | 2 (4)
diarrhea (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 3 (3)
vomiting (Gastrointestinal disorders) | 3 (3)
thromboembolism (vascular access-related) (Vascular disorders) | 1 (1)
enteritis, small bowel (Gastrointestinal disorders) | 1 (1)
edema, facial (General disorders) | 1 (1)
infection with unknown ANC-urinary tract NOS (Renal and urinary disorders) | 1 (1)
calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
hydrocephalus (Nervous system disorders) | 1 (1)
pain-headache (Nervous system disorders) | 1 (1)
ventricular tachycardia (Cardiac disorders) | 1 (1)
pain-right-sided thorax (non-cardiac) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 2 (3)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | RAD001 and Cisplatin and Paclitaxel (N=55)
albumin, serum-low (Metabolism and nutrition disorders) | 7 (8)
alkaline phosphatase (Investigations) | 23 (51)
allergic reaction\hypersensitivity (including drug fever) (Immune system disorders) | 3 (4)
allergy/immunology-other (Immune system disorders) | 3 (3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 22 (44)
anorexia (Metabolism and nutrition disorders) | 12 (18)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 14 (18)
calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 5 (7)
cholesterol, serum-high (hypercholesteremia (Investigations) | 17 (26)
constipation (Gastrointestinal disorders) | 18 (21)
constitutional symptoms-other (General disorders) | 19 (162)
cough (Respiratory, thoracic and mediastinal disorders) | 11 (12)
creatinine (Investigations) | 4 (9)
dermatology/skin-other (Skin and subcutaneous tissue disorders) | 13 (21)
diarrhea (Gastrointestinal disorders) | 20 (28)
dizziness (Gastrointestinal disorders) | 6 (6)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
edema limb (General disorders) | 11 (17)
fatigue (General disorders) | 32 (45)
gastrointestinal-other (Gastrointestinal disorders) | 7 (9)
glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 33 (76)
hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 8 (9)
heartburn/dyspepsia (Gastrointestinal disorders) | 3 (3)
hemoglobin (Blood and lymphatic system disorders) | 52 (182)
hemorrhage, pumonary/upper respiratory-nose (Respiratory, thoracic and mediastinal disorders) | 5 (5)
infection-other (Infections and infestations) | 11 (11)
infection with normal ANC or grade 1 or 2 neutrophils-urinary tract NOS (Renal and urinary disorders) | 3 (3)
insomnia (Psychiatric disorders) | 9 (11)
leukocytes (total WBC) (Blood and lymphatic system disorders) | 33 (141)
nausea (Gastrointestinal disorders) | 34 (44)
neurology-other (Nervous system disorders) | 12 (28)
neuropathy-sensory (Nervous system disorders) | 16 (29)
neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 28 (77)
pain back (Musculoskeletal and connective tissue disorders) | 3 (4)
pain-breast (Reproductive system and breast disorders) | 3 (4)
pain-chest wall (Musculoskeletal and connective tissue disorders) | 3 (3)
pain-extremity-limb (Musculoskeletal and connective tissue disorders) | 4 (6)
pain-head/headache (Nervous system disorders) | 11 (12)
pain-other (General disorders) | 22 (34)
platelets (Blood and lymphatic system disorders) | 39 (85)
potassium-serum-low (hypokalemia) (Metabolism and nutrition disorders) | 20 (33)
pulmonary/upper respiratory-other (Respiratory, thoracic and mediastinal disorders) | 7 (9)
rash acne/acneiform (Skin and subcutaneous tissue disorders) | 7 (8)
sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 14 (25)
taste alteration (dysgeusia) (Nervous system disorders) | 6 (7)
tinnitus (Ear and labyrinth disorders) | 3 (3)
triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 15 (17)
vomiting (Gastrointestinal disorders) | 12 (18)
pain-joint (Musculoskeletal and connective tissue disorders) | 3 (3)
magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 8/52 (11)
metabolic/laboratory-other (Metabolism and nutrition disorders) | 19 (145)
blood/bone marrow-other (Blood and lymphatic system disorders) | 4 (10)
calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 14 (30)
potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (4)
mucositis/stomatitis (clinical exam)-oral cavity (Gastrointestinal disorders) | 10 (12)
mucositis/stomatitis (functional/symptomatic)-oral cavity (Gastrointestinal disorders) | 6 (6)
nail changes (Skin and subcutaneous tissue disorders) | 4 (4)
pruritis/itching (Skin and subcutaneous tissue disorders) | 3 (3)
rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (4)
depression (Psychiatric disorders) | 3 (3)
infection with normal ANC or Grade 1 or 2 neutrophils-nails (Infections and infestations) | 3 (4)
infection with normal ANC or Grade 1 or 2 neutrophils-upper airway NOS (Infections and infestations) | 5 (6)
lymphatics-other (Blood and lymphatic system disorders) | 3 (3)
Pain-neck (Musculoskeletal and connective tissue disorders) | 3 (4)
pain-abdomen NOS (Gastrointestinal disorders) | 4 (5)

LIMITATIONS AND CAVEATS:
All patients began at the same dose level of the study drugs with no de-escalation of dose, thus results were combined for outcomes measures 3, 4, 5, and 6 for Phase II.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes